CLINICAL TRIAL: NCT03058809
Title: Evaluation of the Saftey and Efficacy of the Viatar™ Oncopheresis System in Removing Circulating Tumor Cells From Whole Blood
Brief Title: Evaluation of Viatar™ Oncopheresis System in Removing CTC From Whole Blood
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Viatar LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T30-0002
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Subjects will be their own controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Metastatic Breast, Colon and Prostate Cancer (Experimental): Metastatic breast, colon or prostate cancer patients will have their CTC levels determined on 3 days before treatment with the Viatar Oncopheresis System to establish a baseline value, a pretreatment value, a post treatment value and on 4 additional instances over a period of 7 days post treatment to establish a CTC rebound profile using a validated CTC enumeration system.
  Interventions: Device: Oncopheresis

INTERVENTIONS:
Device: Oncopheresis — Oncopheresis is a type of apheresis incorporating an extracorporeal blood circuit and a filter to separate circulating tumor cells from normal blood components.

SUMMARY:
This study will access the safety and efficacy of the Viatar™ Oncopheresis System to remove a meaningful quantity of circulating tumor cells from the blood of subjects' with breast, colon or prostate solid tumor cancers in a single treatment. CTC reduction will be measured as the change in circulating tumor cells as determined before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of breast, colon or prostate cancer
* No prior cancer therapy or failed first line therapy
* >= 25 CTC per 7.5 mL of blood within 1 week prior to oncopheresis treatment
* > 1 month life expectancy
* Adequate baseline hematological function as assessed by the following laboratory values:

  * Hemoglobin > 9 g/dl
  * Platelets > 100,000/mm3
  * WBC > 3,000/mm3
  * Absolute Neutrophil Count > 1,500/mm3

Exclusion Criteria:

* Coagulation disorders and/or a history of thromboembolic complications, including known hypersensitivity to citrate: e.g., abnormal platelet count, prothrombin time and partial activated thromboplastin time and with a history of deep vein thrombus or pulmonary embolism
* Patients with known immunodeficiency virus (HIV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in Circulating Tumor Cells | % change will be determined on the day of treatment
  % change in enumerated circulating tumor cells after treatment with Viatar Oncopheresis System

SECONDARY OUTCOMES:
Immune system activation | Immune system activation biomarkers will be followed for 7 days post treatment
  To assess the effect of oncopheresis on immune system activation

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Murray, MD, Principal Investigator — Hospital de Carabineros

IPD SHARING:
Plan to Share IPD: Undecided